CLINICAL TRIAL: NCT02694718
Title: A Phase II Study of Capecitabine Plus Oxaliplatin in Combination With Pre-operative Pelvic Radiotherapy in Rectal Cancer
Brief Title: A Study of Capecitabine Plus Oxaliplatin in Combination With Pre-operative Pelvic Radiotherapy in Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Sanofi-Synthélabo (Schweiz) AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18280
Record Dates: First submitted 2016-02-25; First posted 2016-02-29 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

ARMS (1):
- Capecitabine+Oxaliplatin (Experimental): Eligible participants received capecitabine 1000 milligrams per square meter (mg/m^2) on Days 1-14, and 825 mg/m^2 on Days 22-35 and 43-56 twice a day (bid) orally, along with oxaliplatin as a 2-hour intravenous (iv) infusion of 130 mg/m^2/once a day (d) on Day 1 and 50 mg/m^2/d on Days 22, 29, 43 and 50 prior to radiotherapy. Participants received radiation therapy having a fraction dose of 1.8 gray (Gy)/day, 5 days a week, for five consecutive weeks starting on Day 22 of the treatment period. Participants, who completed the treatment period, underwent surgery at Week 14.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is available as 50 mg and 500 mg tablets. It will be administered as a 1000mg/m^2 bid orally on Days 1-14, and at a dose of 825mg/m^2 bid on Days 22-35 and 43-56.
  Other Names: Xeloda, Ro09-1978
Drug: Oxaliplatin — Oxaliplatin is available in vials containing 50 mg or 100 mg. It will be administered as a oxaliplatin 130mg/m^2/d intravenously on Day 1 and 50mg/m^2/d on Days 22, 29, 43 and 50 prior to radiotherapy up to Week 9 followed by surgery period.
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to determine the pathological complete tumor response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced T3/T4 rectal carcinoma with or without nodal involvement requiring surgery of the primary tumor
* Eastern Cooperative Oncology Group performance status 0-2
* Adequate values of laboratory parameters

Exclusion Criteria:

* Evidence of distant metastases
* Previous Chemotherapy or immunotherapy for colorectal cancer
* Previous radiotherapy to the pelvis
* Pre-existing condition which would deter radiotherapy
* Malignancy within last 5 years, except cured basal cell cancer of the skin and in situ cancer of the cervix
* Clinically significant cardiac disease or myocardial infarction within the last 12 months
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome
* Organ allografts
* Concomitant treatment with brivudine, lamivudine, ribavirin or any other nucleoside analogues
* Dihydropyrimidine dehydrogenase (DPD) deficiency
* History of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for oral drug intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03; Primary Completion 2006-08 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (5):
- Switzerland (5):
  - Basel
  - Chur
  - Lucerne
  - Sankt Gallen
  - Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 participants were enrolled in this study conducted from 30 March 2005 to 28 November 2006 at 6 centers in Switzerland.
Groups:
- Capecitabine + Oxaliplatin: Eligible participants received capecitabine 1000 milligrams per square meter (mg/m^2) on Days 1-14, and 825 mg/m^2 on Days 22-35 and 43-56 twice a day (bid) orally, along with oxaliplatin as a 2-hour intravenous (iv) infusion of 130 mg/m^2/once a day (d) on Day 1 and 50 mg/m^2/d on Days 22, 29, 43 and 50 prior to radiotherapy. Participants received radiation therapy having a fraction dose of 1.8 gray (Gy)/day, 5 days a week, for five consecutive weeks starting on Day 22 of the treatment period. Participants, who completed the treatment period, underwent surgery at Week 14.
Period: Overall Study
Arm/Group | Capecitabine + Oxaliplatin
Started | 60
Completed | 58
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who received at least one dose of any of the study treatments and who had a baseline assessment.
Groups:
- Capecitabine + Oxaliplatin: Eligible participants received capecitabine 1000 mg/m^2 on Days 1-14, and 825 mg/m^2 on Days 22-35 and 43-56 bid orally, along with oxaliplatin as a 2-hour iv infusion of 130 mg/m^2/once a day (d) on Day 1 and 50 mg/m^2/d on Days 22, 29, 43 and 50 prior to radiotherapy. Participants received radiation therapy having a fraction dose of 1.8 Gy/day, 5 days a week, for five consecutive weeks starting on Day 22 of the treatment period. Participants, who completed the treatment period, underwent surgery at Week 14.
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Tumor Response
Description: Pathological complete tumor response was defined as grade 3 or 4 in the histological grading of regression according to Dworak classification. Grade 0 is no regression; Grade 1 is dominant tumor mass with obvious fibrosis and/or vasculopathy; Grade 2 is dominantly fibrotic changes with few tumor cells or groups; Grade 3 is defined as very few (difficult to find microscopically) tumor cells in fibrotic tissue with or without mucous substance; Grade 4 is defined as no tumor cells, only fibrotic mass (total regression or response).
Time Frame: Up to Week 16
Population: The intent to treat (ITT) population included all participants, who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 60
Percentage of participants | 23 [13.4 to 36.0]

2. Secondary Outcome: Percentage of Participants With Sphincter-preservation
Description: Percentage of participants with sphincter-preservation is reported.
Time Frame: Up to Week 16
Population: ITT population included all participants, who received at least one dose of study drug. Two participants from the ITT population did not undergo surgery (one died, one withdrew consent).
Measure: Number; unit: Percentage of participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 58
Percentage of participants | 84.48

3. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Number of participants with marked laboratory abnormalities is reported.
Time Frame: Up to Week 16
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 60
Participants
  Hemoglobin | 7
  Hematocrit | 7
  Erythrocytes | 16
  Leucocytes total | 8
  Neutrophils | 9
  Basophils | 1
  Eosinophils | 2
  Monocytes | 2
  Lymphocytes | 42
  Platelets | 13
  ASAT/SGOT | 2
  ALAT/SGPT | 10
  Serum albumin | 3
  Total protein | 2
  Serum creatinine | 2
  Glucose | 13
  Sodium | 2
  Potassium | 2
  Calcium | 2

4. Secondary Outcome: Percentage of Participants With Resection (R0) in Participants With T4 Rectal Cancer
Description: R0 resection was defined as complete resection of the tumor with adequate tumor-free margins and regional lymph node extirpation as confirmed by pathology after pre-operative chemotherapy plus capecitabine + oxaliplatin therapy.
Time Frame: Up to Week 16
Population: The ITT consists of all included participants, who received at least one dose of study drug. Five participants from ITT population with T4 rectal cancer underwent surgery.
Measure: Number; unit: Percentage of participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 5
Percentage of participants | 100

5. Secondary Outcome: Percentage of Participants With Downstaging of Primary Tumor and/or Lymph Nodes
Description: Downstaging of primary tumor (T) and/or lymph nodes (N) was defined as decrease by 1 point in T-value and/or N-value (comparing at screening and after treatment). It was assessed by colonoscopy, pathology, endosonography of rectum, chest X-ray, abdominopelvic Computed Tomography and Magnetic Resonance Imaging. Staging for tumor are: TX (primary tumor cannot be assessed), T0 (no evidence of primary tumor), Tis (carcinoma in situ), T1 (tumor invades submucosa), T2 (tumor invades muscularis propria), T3 (tumor invades through muscularis propria into subserosa/into non-peritonealized pericolic/perirectal tissues, T4 (tumor directly invades other organs or structures). Staging for lymph nodes are: NX (regional lymph nodes cannot be assessed), N0 (no regional lymph node metastasis), N1 (metastasis in 1 to 3 regional lymph nodes), N2 (metastasis in 4 or more regional lymph nodes).
Time Frame: From screening to Week 16
Population: ITT population included all participants, who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 60
Percentage of participants
  T stage | 47
  N stage | 48
  Overall | 65

6. Secondary Outcome: Percentage of Participants With Pathological Incomplete Tumor Response
Description: Pathological incomplete tumor response was defined as grade 1 or 2 in the histological grading of regression according to Dworak grading of regression. Pathological incomplete tumor response rate, Grade 1: dominant tumor mass with obvious fibrosis and/or vasculopathy; Grade 2: dominantly fibrotic changes with few tumor cells or groups (easy to find) were assessed.
Time Frame: Up to Week 16
Population: ITT population included all participants, who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 60
Percentage of participants | 72 [58.6 to 82.5]

7. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in participants or clinical investigation participants administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 16
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 60
Participants
  Any AEs | 59
  Any SAEs | 8

ADVERSE EVENTS:
Time Frame: Up to Week 16
Description: AE is defined as any untoward medical occurrence in participants or clinical investigation participants administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. A SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalisation or prolongation of hospitalisation or results in disability/incapacity, and congenital anomaly/birth defect.
Arm/Group | Capecitabine + Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 8/60
Other Adverse Events (participants affected / at risk) | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin (N=60)
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 1
Anal Haemorrhage (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin (N=60)
Diarrhoea (Gastrointestinal disorders) | 42
Nausea (Gastrointestinal disorders) | 20
Proctitis (Gastrointestinal disorders) | 14
Abdominal Pain (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Painful Defaecation (Gastrointestinal disorders) | 7
Proctalgia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 27
Temperature Intorlerance (General disorders) | 4
Pain (General disorders) | 3
Weight Decrease (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 11
Neuropathy (Nervous system disorders) | 13
Paraesthesia (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 5
Peripheral Sensory Neropathy (Nervous system disorders) | 5
Neuropathy Peripheral (Nervous system disorders) | 4
Pollakiuria (Renal and urinary disorders) | 12
Dysuria (Renal and urinary disorders) | 5
Nocturia (Renal and urinary disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hand and Foot Syndrome (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.